CLINICAL TRIAL: NCT03157895
Title: A Trial of Connecting to Prevent Drug Abuse and Risky Behavior in Foster Teens
Brief Title: A Trial of Connecting to Promote Foster Teen Well-Being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Alliance for Child Welfare Excellence (Unknown); Washington State Department of Social and Health Services (Other)
Responsible Party: Principal Investigator, Kevin Haggerty, Director, Social Development Research Group, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D012912S
Record Dates: First submitted 2017-04-27; First posted 2017-05-17 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Relationship, Family (Foster); Substance Use Prevention
Keywords: Foster Families

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Interviewers should be blind to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program group (Experimental): This group receives the Connecting program with telephone support. It's anticipated the program will take up to 14 weeks to complete.
  Interventions: Behavioral: Connecting
- Comparison group (No Intervention): This group receives Children's Administration services as usual.

INTERVENTIONS:
Behavioral: Connecting — Connecting was adapted for use within the child welfare system from the Staying Connected With Your Teen program that has been demonstrated to prevent substance abuse, risky sexual behavior, and violence during adolescence.
  Other Names: Staying Connected With Your Teen
  Arms: Program group

SUMMARY:
This study evaluates the efficacy of a self-directed parenting program called Connecting in reducing risk of substance use and other risky behaviors in young foster teens (ages 11-15). Half of the participants will receive services as usual from the foster system, while half will participate in the Connecting program. Connecting is a 10-week, self-directed parenting workbook with two digital video discs (DVDs). Families receive weekly telephone support as they complete the program.

ELIGIBILITY:
Inclusion Criteria:

* Foster youth ages 11-15 years
* In current placement 60+ days
* In relative/suitable adult care, in licensed relative/suitable adult care, in licensed foster care, in dependency guardianship
* Caregiver and teen speak English well enough to use the program manual and respond to survey questions

Exclusion Criteria:

* The teen has regularly used drugs or alcohol in the last 30 days
* The teen has been involved in the criminal justice system
* The placement is not viewed as stable
* The caregiver is not committed to a long-term placement
* The teen will not likely be in the placement for at least 6 months
* Group home placements and behavioral rehabilitative services placements

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Delay in drug use initiation | 2 year follow up
  Monitoring the Future (Johnston et al., 2002). Communities that Care Youth Survey (CTC) (Hawkins & Catalano, 2004).
Substance use frequency | 2 year follow up
  Monitoring the Future (Johnston et al., 2002). Communities that Care Youth Survey (Hawkins & Catalano, 2004).
Non-violent delinquent behavior frequency | 2 year follow up
  Seattle Social Development Project (SSDP) (Hawkins et al., 1999). Raising Healthy Children (Catalano et al., 2005).
Violent delinquent behavior frequency | 2 year follow up
  Seattle Social Development Project (Hawkins et al., 1999).
Delay in initiation of sexual activity | 2 year follow up
  National Longitudinal Survey of Youth (Center for Human Research, 2003). Sexual Risk and Behavior Attitudes and Self Efficacy Scale (Basen Enquist et al., 1996). Communities that Care Youth Survey (Hawkins & Catalano, 2004).

SECONDARY OUTCOMES:
Residential placement stability | 2 year follow up
  Child Welfare Administrative Data
Growth in caregiver/youth bonding | 1 and 2 year follow up
  Communities that Care Youth Survey (Hawkins & Catalano, 2004). Armsden & Greenberg (1987).
Youth attitudes about HIV related risks | 1 and 2 year follow up
  Sexual Risk and Behavior Attitudes and Self Efficacy Scale (Basen Enquist et al.,1996)
Youth attitudes favorable toward substance use | 1 and 2 year follow up
  Communities that Care Youth Survey (Hawkins & Catalano, 2004)

OTHER OUTCOMES:
Opportunities for prosocial involvement in the family | 1 and 2 year follow up
  Alabama Parenting Questionnaire (Shelton et al., 1999)
Problem solving skills (youth) | 1 and 2 year follow up
  Raising Healthy Children (Catalano et al., 2005)
Refusal skills (youth) | 1 and 2 year follow up
  Seattle Social Development Project (1999)
Children's coping | 1 and 2 year follow up
  University of Washington Parenting Clinic (2001)
Rewards and recognition in the family scale | 1 and 2 year follow up
  Raising Healthy Children (Catalano et al., 2005)
Change in family guidelines | 1 and 2 year follow up
  Alabama Parenting Questionnaire (1999)
Change in caregiver monitoring | 1 and 2 year follow up
  Parental Monitoring; Kerr and Stattin (2000). Raising Healthy Children monitoring scale (Catalano et al., 2005).
Change in inconsistent discipline and consequences | 1 and 2 year follow up
  Alabama Parenting Questionnaire (Shelton et al., 1999)

CONTACTS AND LOCATIONS:
Locations (1):
- The Social Development Research Group, University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haggerty KP, Barkan SE, Skinner M, Ben Packard W, Cole JJ. Feasibility of Connecting, a Substance-Abuse Prevention Program for Foster Teens and their Caregivers. J Soc Social Work Res. 2016 Winter;7(4):639-659. doi: 10.1086/686986. Epub 2016 Oct 18. PMID 27891209
- [Background] Barkan SE, Salazar AM, Estep K, Mattos LM, Eichenlaub C, Haggerty KP. Adapting an evidence based parenting program for child welfare involved teens and their caregivers. Child Youth Serv Rev. 2014 Jun;41:53-61. doi: 10.1016/j.childyouth.2014.03.006. PMID 26052172
- [Background] Storer HL, Barkan SE, Stenhouse LL, Eichenlaub C, Mallillin A, Haggerty KP. In search of connection: The foster youth and caregiver relationship. Child Youth Serv Rev. 2014 Jul;42:110-117. doi: 10.1016/j.childyouth.2014.04.008. PMID 26052173
- [Background] Storer HL, Barkan SE, Sherman EL, Haggerty KP, Mattos LM. Promoting Relationship Building and Connection: Adapting an Evidence-Based Parenting Program for Families Involved in the Child Welfare System. Child Youth Serv Rev. 2012 Sep 1;34(9):10.1016/j.childyouth.2012.05.017. doi: 10.1016/j.childyouth.2012.05.017. PMID 24347754
- [Background] Salazar AM, McCowan KJ, Cole JJ, Skinner ML, Noell BR, Colito JM, Haggerty KP, Barkan SE. Developing Relationship-Building Tools for Foster Families Caring for Teens who are LGBTQ2S. Child Welfare. 2018;96(2):75-97. PMID 29861503
- [Derived] Haggerty KP, Barkan SE, Caouette JD, Skinner ML, Hanson KG. Two-Year Risk Behavior Outcomes from Connecting, a Prevention Program for Caregivers and Youth in Foster Care. Prev Sci. 2023 Jan;24(1):15-26. doi: 10.1007/s11121-022-01390-4. Epub 2022 Jul 4. PMID 35788868